CLINICAL TRIAL: NCT02436005
Title: Dispensing Study for the Phenacite Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-15-16
Record Dates: First submitted 2015-05-01; First posted 2015-05-06 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Phenacite (Experimental): Subjects will be randomized to wear the Phenacite contact lenses binocularly.
  Interventions: Device: Phenacite; Device: comfilcon A
- comfilcon A (Active Comparator): Subjects will be randomized to wear the comfilcon A contact lenses binocularly.
  Interventions: Device: Phenacite; Device: comfilcon A

INTERVENTIONS:
Device: Phenacite — Subjects will be randomized to wear the Phenacite contact lenses binocularly.
Device: comfilcon A — Subjects will be randomized to wear the comfilcon A contact lenses binocularly.

SUMMARY:
Dispensing Study for the Phenacite Project.

The investigational test lens was not the final optical design and the study was not used for design validation.

DETAILED DESCRIPTION:
Evaluate the objective and patient-reported visual acceptability of the Phenacite contact lens.

ELIGIBILITY:
Inclusion Criteria:

* Oculo-visual examination in the last two years
* Between 18 and 35 years of age and has full legal capacity to volunteer
* Has read and understood the informed consent letter
* Is willing and able to follow instructions and maintain the appointment schedule
* Is correctable to a visual acuity of 20/25 or better (in each eye) with their habitual correction or 20/20 best corrected
* Currently wears, or has previously successfully worn, soft contact lenses between -1.00D and -4.00D
* Spherical Contact Lens Rx between -1.00 and -4.00 and spectacle cylinder ≤-0.75
* Has not worn lenses for at least 12 hours before the initial visit
* Has a subjective response at baseline, which indicates suitability for this study
* Currently spends a minimum of 4 hours a day; 5 days a week on digital devices and can replicate this time during the study period
* Is willing and able to wear the study contact lenses a minimum of 10 hours per day; 5 days a week.

Exclusion Criteria:

* Has never worn contact lenses before
* Any systemic disease affecting ocular health
* Is using any systemic or topical medications that will affect ocular health
* Has known sensitivity to the diagnostic pharmaceuticals or study products used in this study.
* Has any ocular pathology or anomaly that would affect the wearing of the lenses
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye
* Is aphakic
* Has anisometropia of >1.00
* Has undergone corneal refractive surgery
* Has strabismus
* Has any ocular amblyopia >= 1line of HC Visual Acuity
* Is participating in any other type of eye related clinical or research study
* Has participated in study CV-14-32.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pete Kollbaun, OD PhD, Principal Investigator — CORL Indiana University
Locations (1):
- Clinical Optics Research Lab (CORL) Indiana University School of Optometry, Indiana University, Bloomington, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phenacite Then Comfilcon A: Subjects will be randomized to wear the Phenacite contact lenses binocularly for two weeks then cross-over to comfilcon A lenses for two weeks.
  Phenacite: contact lenses comfilcon A: Contact Lenses
- Comfilcon A Then Phenacite: Subjects will be randomized to wear comfilcon A contact lenses for two weeks then cross-over to Phenacite Lenses for two weeks.
  comfilcon A: Contact Lenses Phenacite : Contact Lenses
Period: First Intervention
Arm/Group | Phenacite Then Comfilcon A | Comfilcon A Then Phenacite
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Phenacite Then Comfilcon A | Comfilcon A Then Phenacite
Started | 12 | 13
Completed | 12 | 12
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects will be randomized to wear the Phenacite and comfilcon A contact lenses binocularly for two weeks.
  Phenacite: contact lenses (Not the final Design - Further clinical studies were conducted to validate the new design)
  comfilcon A: contact lenses
Arm/Group | Overall Study
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Subjective Ratings of Lens Comfort
Description: Subjective ratings of lens comfort. Comfort Scale (0,100; 0=extremely uncomfortable/cannot tolerate; 100 = extremely comfortable/cannot be felt)
Time Frame: Baseline (after 15 minutes of lens dispense)
Population: One subject was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Phenacite: Subjects will be randomized to wear the Phenacite contact lenses binocularly.
  Phenacite: contact lenses
- Comfilcon A: Subjects will be randomized to wear the comfilcon A contact lenses binocularly.
  comfilcon A: contact lenses
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
units on a scale | 86.50 (14.99) | 90.13 (8.60)

2. Primary Outcome: Subjective Ratings of Lens Comfort
Description: as for outcome 1
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
units on a scale | 66.46 (25.22) | 71.71 (24.62)

3. Primary Outcome: Over Refraction for Optimized Distance Acuity
Description: Over Refraction for optimized distance acuity measured using logMAR
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
logMAR
  OD (oculus dexter - right eye) | -0.10 (0.09) | 0.00 (0.00)
  OS (Oculus sinister - left eye) | -0.02 (0.07) | 0.00 (0.00)

4. Primary Outcome: Binocular Distance Visual Acuity - High Illumination High Contrast
Description: Binocular Distance Visual Acuity - High Illumination High Contrast was measured using logMAR
Time Frame: Baseline (after 5 minutes of lens dispense)
Population: One subject was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
logMAR | -0.18 (0.06) | -0.21 (0.06)

5. Primary Outcome: Binocular Distance Visual Acuity - High Illumination High Contrast
Description: Binocular Distance Visual Acuity - High Illumination High Contrast was measured using logMAR
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
logMAR | -0.19 (0.07) | -0.20 (0.05)

6. Primary Outcome: Binocular Distance Visual Acuity - Low Illumination High Contrast
Description: Binocular Distance Visual Acuity - Low Illumination High Contrast was measured using logMAR
Time Frame: Baseline (after 5 minutes of lens dispense)
Population: One subject was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
logMAR | 0.03 (0.08) | 0.00 (0.07)

7. Primary Outcome: Binocular Distance Visual Acuity - Low Illumination High Contrast
Description: Binocular Distance Visual Acuity - Low Illumination High Contrast was measured using logMAR
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
logMAR | 0.00 (0.09) | 0.00 (0.06)

8. Primary Outcome: Binocular Near Visual Acuity - High Illumination High Contrast
Description: Binocular Near Visual Acuity - High Illumination High Contrast was measured using logMAR
Time Frame: Baseline (after 5 minutes of lens dispense)
Population: One subject was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
logMAR | -0.16 (0.06) | -0.19 (0.06)

9. Primary Outcome: Binocular Near Visual Acuity - High Illumination High Contrast
Description: Binocular Near Visual Acuity - High Illumination High Contrast was measured using logMAR
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
logMAR | -0.20 (0.06) | -0.18 (0.06)

10. Primary Outcome: Binocular Near Visual Acuity - Low Illumination High Contrast
Description: Binocular Near Visual Acuity - Low Illumination High Contrast was measured using logMAR
Time Frame: Baseline (after 5 minutes of lens dispense)
Population: One subject was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
logMAR | 0.01 (0.07) | -0.01 (0.10)

11. Primary Outcome: Binocular Near Visual Acuity - Low Illumination High Contrast
Description: Binocular Near Visual Acuity - Low Illumination High Contrast was measured using logMAR
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
logMAR | -0.02 (0.09) | -0.03 (0.08)

12. Secondary Outcome: Lens Fit - Post Blink Movement
Description: Investigator assessment of Amount of movement (to the nearest 0.1mm) immediately after the blink (0.1mm steps)
Time Frame: Baseline (after 15 minutes of lens dispense)
Population: One Subject was excluded from the analysis
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
mm
  OD (oculus dexter - right eye) | 0.23 (0.07) | 0.20 (0.06)
  OS(oculus sinister - left eye) | 0.23 (0.07) | 0.22 (0.07)

13. Secondary Outcome: Lens Fit - Post Blink Movement
Description: Investigator assessment of Amount of movement (to the nearest 0.1mm) immediately after the blink (0.1mm steps)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
mm
  OD (oculus dexter - right eye) | 0.24 (0.09) | 0.23 (0.08)
  OS (oculus sinister - left eye) | 0.25 (0.08) | 0.24 (0.07)

14. Secondary Outcome: Push - Up Test for Lens Tightness
Description: Investigator assessment using Continuous Scale 0-100% (1% steps): 0%=Falls from cornea without lid support, 50%=Optimum, 100%=No movement
Time Frame: Baseline (after 15 minutes of lens dispense)
Population: One Subject was excluded from the analysis
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
mm
  OD (oculus Dexter - Right eye) | 50.43 (5.09) | 51.52 (5.40)
  OS (Oculus Sinister - Left eye) | 49.78 (4.77) | 50.65 (4.73)

15. Secondary Outcome: Push - Up Test for Lens Tightness
Description: as for outcome 14
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
mm
  OD (oculus dexter - right eye) | 52.83 (7.64) | 49.35 (4.50)
  OS (Oculus Sinister - Left Eye) | 51.30 (5.94) | 48.70 (4.23)

16. Secondary Outcome: Lens Mobility Rating
Description: Investigator assessment using 5 Categories in 0.50 steps: 0=Immobile - no lag in any versions, 1=Restricted - no lag in some directions but slight lag (0-0.25mm) in others, 2=Secure - slight lag (0.25-0.5mm in each version), 3=Unrestricted - freely lags in a controlled manner on all versions, but not excessive (0.5-1.0mm), 4=Very mobile - excessive lag (>1mm) on versions in all directions in 0.25 steps
Time Frame: Baseline (after 15 minutes of lens dispense)
Population: One Subject was excluded from the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
units on a scale
  OD (oculus dexter - Right Eye) | 3.07 (0.34) | 2.99 (0.36)
  OS (Oculus Sinister - Left eye) | 3.09 (0.32) | 3.01 (0.35)

17. Secondary Outcome: Lens Mobility Rating
Description: as for outcome 16
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
units on a scale
  OD (oculus dexter - right eye) | 2.91 (0.35) | 3.08 (0.31)
  OS (oculus sinister - left eye) | 3.00 (0.33) | 3.10 (0.28)

18. Secondary Outcome: Overall Lens Fit Acceptance
Description: Investigator assessment using 5 Categories in 0.25 steps: 0=Can't be worn, 1=Poor - should not be dispensed although no immediate danger, 2=Fair, 3=Good, 4=Optimum in 0.25 steps
Time Frame: Baseline (after 15 minutes of lens dispense)
Population: One Subject was excluded from the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
units on a scale
  OD (oculus dexter - right eye) | 3.35 (0.25) | 3.30 (0.32)
  OS ( oculus sinister - Left Eye) | 3.37 (0.24) | 3.30 (0.28)

19. Secondary Outcome: Overall Lens Fit Acceptance
Description: as for outcome 18
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
units on a scale
  OD (oculus dexter- right eye) | 3.25 (0.35) | 3.34 (0.34)
  OS (oculus sinister - left eye) | 3.32 (0.32) | 3.36 (0.36)

20. Secondary Outcome: Subjective Ratings for Vision Quality - Distance Vision
Description: Patient subjective scoring using 0-100 continuous scale for Distance Quality of Vision: 0=extremely poor vision all of the time. Cannot function; 20= Frequently annoying vision problems; 40=Occasionally annoying vision problems; 60=occasionally noticeable but not annoying vision problems; 80=rarely noticeable vision problems; 100=excellent vision all of the time
Time Frame: Baseline (after 15 minutes of lens dispense)
Population: One Subject was excluded from the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
units on a scale | 86.58 (17.13) | 91.3 (10.64)

21. Secondary Outcome: Subjective Ratings for Vision Quality - Distance Vision
Description: as for outcome 20
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
units on a scale | 85.33 (20.5) | 88.88 (15.34)

22. Secondary Outcome: Subjective Ratings for Vision Quality - Near Vision
Description: Patient subjective scoring using 0-100 continuous scale for Near Quality of Vision: 0=extremely poor vision all of the time. Cannot function; 20= Frequently annoying vision problems; 40=Occasionally annoying vision problems; 60=occasionally noticeable but not annoying vision problems; 80=rarely noticeable vision problems; 100=excellent vision all of the time
Time Frame: Baseline (after 15 minutes of lens dispense)
Population: One Subject was excluded from the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
units on a scale | 92.00 (11.16) | 92.63 (7.70)

23. Secondary Outcome: Subjective Ratings for Vision Quality - Near Vision
Description: as for outcome 22
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
units on a scale | 84.83 (23.88) | 85.88 (21.67)

24. Secondary Outcome: Subjective Ratings for Vision Quality - Computer Vision
Description: Patient subjective scoring using 0-100 continuous scale for Computer Vision: 0=extremely poor vision all of the time. Cannot function; 20= Frequently annoying vision problems; 40=Occasionally annoying vision problems; 60=occasionally noticeable but not annoying vision problems; 80=rarely noticeable vision problems; 100=excellent vision all of the time
Time Frame: Baseline (after 15 minutes of lens dispense)
Population: One Subject was excluded from the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
units on a scale | 92.79 (10.75) | 93.17 (8.91)

25. Secondary Outcome: Subjective Ratings for Vision Quality - Computer Vision
Description: as for outcome 24
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
units on a scale | 85.04 (21.27) | 89.08 (15.06)

26. Secondary Outcome: Subjective Ratings for Vision Quality - Overall Vision
Description: Patient subjective scoring using 0-100 continuous scale for Overall Vision: 0=extremely poor vision all of the time. Cannot function; 20= Frequently annoying vision problems; 40=Occasionally annoying vision problems; 60=occasionally noticeable but not annoying vision problems; 80=rarely noticeable vision problems; 100=excellent vision all of the time
Time Frame: Baseline (after 15 minutes of lens dispense)
Population: One Subject was excluded from the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
units on a scale | 91.00 (10.64) | 92.67 (7.41)

27. Secondary Outcome: Subjective Ratings for Vision Quality - Overall Vision
Description: as for outcome 26
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
units on a scale | 85.96 (17.66) | 88.63 (14.36)

28. Secondary Outcome: Corneal Staining Extent
Description: Corneal staining extent was assessed on a scale of 0-4 (0-No Staining, 1 - 1-15% of area, 2- 16-30% of area, 3- 31-45% of area, 4- >45% of area
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
units on a scale
  Central | 0.02 (0.14) | 0.00 (0.00)
  Nasal | 0.00 (0.00) | 0.00 (0.00)
  Temporal | 0.00 (0.00) | 0.00 (0.00)
  Superior | 0.00 (0.00) | 0.04 (0.20)
  Inferior | 0.21 (0.50) | 0.42 (0.58)

29. Secondary Outcome: Conjunctival Staining
Description: Conjunctival staining was assessed on a scale of 0-4, 0.50 steps (0-None, 1 - Minimal diffuse punctuate, 2- Coalescent Punctuate, 3- confluent, 4- Deep confluent
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 24 | 24
units on a scale
  Nasal | 0.48 (0.46) | 0.38 (0.57)
  Temporal | 0.11 (0.36) | 0.18 (0.43)
  Superior | 0.00 (0.00) | 0.05 (0.26)
  Inferior | 0.02 (0.10) | 0.10 (0.27)

ADVERSE EVENTS:
Time Frame: From dispense up to two weeks on each study lenses, a total of four weeks.
Groups:
- Phenacite: Subjects will be randomized to wear the Phenacite contact lenses binocularly for two weeks.
  Phenacite: contact lenses
- Comfilcon A: Subjects will be randomized to wear comfilcon A contact lenses binocularly for two weeks.
  comfilcon A: contact lenses binocularly.
Arm/Group | Phenacite | Comfilcon A
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No